CLINICAL TRIAL: NCT01334827
Title: Rational Development of Combination Microbicide Therapies: A Formative Study to Explore the Sensory Perceptions of Vaginal Product Users (Project MIST)
Brief Title: A Formative Study to Explore the Sensory Perceptions of Vaginal Product Users
Acronym: Project-MIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: ImQuest Pharmaceuticals, Inc. (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11800; R33AI076967 (NIH)
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Results first posted 2020-12-08 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Microbicide Delivery System Acceptability
Keywords: topical microbicide; primary prevention; HIV; drug delivery systems
MeSH Terms: interventions — Radiation Dosage; Dyrk Kinases; RID

STUDY DESIGN:
Intervention Model Description: Mixed Methods Measurement Development study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Formulations (Other): high volume gel; low volume gel; vaginal film
  Interventions: Other: high volume gel; Other: low volume gel; Other: vaginal film

INTERVENTIONS:
Other: high volume gel — 4 mL HEC
  Other Names: Gray
Other: low volume gel — 2 mL HEC
  Other Names: Red
Other: vaginal film — 1" x 2" intravaginal quick-dissolving film
  Other Names: Blue

SUMMARY:
The purpose of the study is to compare, contrast, and characterize the range of user perceptions and potential acceptability of three (3) topical vaginal microbicide dosage forms.

DETAILED DESCRIPTION:
The success of microbicide products will derive from the synergy of their biological functionality and user acceptability. Biological functionality is the integrated result of safe and effective anti-HIV compounds incorporated into dosage forms or devices that successfully deliver those compounds to target tissues, fluids, and pathogens. Acceptability is a multi-factorial phenomenon that accounts for the personal, dyadic, product-related, and social contexts that potentiate - or not - a woman's decision to use a microbicide. Acceptability (assessed, in part, by the users' sensory perceptions of products during use) depends strongly upon dosage forms and/or delivery systems with biophysical functions and/or mechanical and materials properties that are most conducive to human use. Without both, microbicides' potential to decisively alter the public health impact of HIV/AIDS and other sexually transmitted infections will be largely limited. The current protocol will specifically study the impact of gel volume on user perceptions, as well as extend user perception scale development to include those properties and product "behaviors" experienced when using a vaginal film.

ELIGIBILITY:
Inclusion Criteria:

Women who:

* are between the ages of 18 and 45
* report vaginal sex with their male sexual partner in the past 6 months
* report being in a monogamous sexual relationship with their male partner
* report consistent use of an effective birth control method: e.g., hormonal contraceptive, IUD, bilateral tubal ligation, Essure® or any non-incisional permanent birth control procedure, hysterectomy (partial or total, with/without oophorectomy), partner's vasectomy/salpingectomy
* are able to tolerate film use, as measured by pelvic exam at Visit 1B
* are willing to refrain from any vaginal product use (inclusive of douching) for 48 hours before Visit 1B and until they complete all study activities (except for study-related products)
* are willing to refrain from having vaginal intercourse 24 hours before Visit 1B and Visits 2-4
* are willing to use condoms for vaginal-penile sex between all study visits (Visits 1A - 4)
* are willing to refrain from any non-penile vaginal penetration during dosage form evaluation visits (Visits 2-4)
* are willing to undergo HIV testing and receive test results and counseling.

Men who:

* are at least 18 years of age
* report vaginal sex with their female sexual partner in the past 6 months
* report being in a monogamous sexual relationship with their female sexual partner
* are willing to refrain from having vaginal intercourse 24 hours before Visit 1B and Visits 2-4
* are willing to use condoms for vaginal-penile sex between all of study visits (Visits 1A-4)
* are willing to refrain from any non-penile vaginal penetration during dosage form evaluation visits (Visits 2-4)
* are willing to use a non-lubricated latex condom (provided) for penile-vaginal intercourse during dosage form evaluation visits (Visits 2-4)
* are willing to undergo HIV testing and receive test results and counseling.

Exclusion Criteria:

Women and men will be ineligible if:

* they are unable or unwilling to give informed consent
* their partner is unable or unwilling to give informed consent
* they are currently enrolled in other vaginal product study/studies
* they are STI (Neisseria gonorrhea, Chlamydia trachomatis, bacterial vaginosis, trichomoniasis, syphilis), HIV positive upon screening (Visit 1A), or pregnant (females) at any study visit
* they are breastfeeding, or have completed menopause (i.e., at least 12 months without menstrual periods) (female participants only)
* they are currently attempting to get pregnant or have an intention to get pregnant during their participation in the study
* they have clinically significant abnormal pelvic findings and/or findings requiring therapy as a function of clinical exam at Visits 1A and/or 1B (female participants only)
* they report being within 30 days of their last pregnancy outcome or gynecologic surgical procedure
* they have known, or suspected, allergies to any component of the study products or similar ingredients in other products
* they have known, or suspected, allergies to latex
* they have any condition that, in the opinion of the study clinician or principle investigator, would compromise the participant´s ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Buckheit, PhD, Principal Investigator — ImQuest Pharmaceuticals; Kathleen Morrow, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited (RI, MA USA) via call-lists, flyers, ads, internet/social media, clinics, CBOs, word-of-mouth.
Groups:
- Female and Male Members of Monogamous Couples: Heterosexual mutually monogamous couples in good general health evaluate 3 topical vaginal formulations (all placebo)
Period: Overall Study
Arm/Group | Female and Male Members of Monogamous Couples
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Female Member of Couple Enrolled; Male Member of Couple Enrolled: Heterosexual mutually monogamous couples in good general health evaluate 3 topical vaginal formulations (all placebo)
- Total: Total of all reporting groups
Arm/Group | Female Member of Couple Enrolled | Male Member of Couple Enrolled | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Customized [Count of Participants; unit: Participants]
  18-29 | 12 | 12 | 24
  30+ | 12 | 12 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 0 | 24
  Male | 0 | 24 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 21 | 22 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 15 | 17 | 32
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 24 | 48
Current Contraceptive Use [Count of Participants; unit: Participants] — Population: Only females assessed
  Participants
    number analyzed (Participants) | 24 | 0 | 24
    Hormonal Contraceptive | 17 |  | 17
    Non-Hormonal Contraceptive | 7 |  | 7
History of STD diagnosis [Count of Participants; unit: Participants] | 4 | 2 | 6
Yearly Income [Count of Participants; unit: Participants]
  Less than $15,000 annually | 12 | 6 | 18
  $15,000-$36,000 annually | 7 | 10 | 17
  More than $36,000 annually | 5 | 8 | 13
Vaginal Deliveries [Count of Participants; unit: Participants] — Population: Only females assessed
  Participants
    number analyzed (Participants) | 24 | 0 | 24
    (all) | 9 |  | 9

OUTCOME MEASURES:

1. Primary Outcome: User Sensory Perception & Experience (USPE; Perceptibility) Scale Item Means
Description: USPE Sum of averaged item means/# items (min:max 1:5); 1=Do not agree at all;2=Agree a little;3=Agree somewhat;4=Agree a lot;5=Agree completely. Products:Low volume gel, high volume gel, film.Initial Penetration:Smoothness/lubricity; Initial Lubrication:Coating/lubricating; Spreading Behavior:Ease of stroke, product spread; Product Awareness:Feel intravaginally during sex (movement, felt betw vaginal wall-penis); Perceived Wetness:Covering entire vagina; as after orgasm; Stimulating: enhanced pleasure; Messiness:Perceptions of watery/messiness; Leakage:Sensations of leaking during/after sex; in pubic hair; need to clean; Pre-coital Leakage:Product felt/leakage noticed on panty liner before sex; Naturalness:Sensation of naturalness; leakage looked like vaginal fluid; Lubricity:Wetness before sex; slipperiness/lubricity during sex; Effortful:Effort needed at penetration; effort difficulty/dryness; Pleasure:Partner's stimulation; Noticeable:Male sensation during sex, messiness, thickness
Time Frame: 4-5 visits over an average of 8-12 weeks
Population: Perceived Pre-Sex Leakage not applicable for Male members of enrolled couples
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Female Members; Male Members: Heterosexual mutually monogamous couples in good general health evaluate 3 topical vaginal formulations (all placebo)
Arm/Group | Female Members | Male Members
Number analyzed (Participants) | 24 | 24
units on a scale
  SEX: Initial Penetration [Low Volume Gel] | 3.64 (1.20) | 3.86 (0.75)
  SEX: Initial Penetration [High Volume Gel] | 4.35 (0.76) | 3.83 (0.74)
  SEX: Initial Penetration [Film] | 1.74 (1.16) | 2.06 (1.03)
  SEX: Initial Lubrication [Low Volume Gel] | 3.54 (1.22) | 3.58 (0.72)
  SEX: Initial Lubrication [High Volume Gel] | 3.89 (1.02) | 3.78 (0.77)
  SEX: Initial Lubrication [Film] | 2.55 (1.27) | 2.60 (1.04)
  SEX: Product Awareness [Low Volume Gel] | 2.55 (0.94) | 2.72 (0.95)
  SEX: Product Awareness [High Volume Gel] | 2.89 (1.10) | 3.10 (1.16)
  SEX: Product Awareness [Film] | 1.73 (0.68) | 2.04 (0.88)
  SEX: Perceived Wetness [Low Volume Gel] | 2.88 (1.33) | 3.00 (0.91)
  SEX: Perceived Wetness [High Volume Gel] | 3.43 (0.95) | 3.38 (1.04)
  SEX: Perceived Wetness [Film] | 1.74 (0.85) | 1.94 (0.86)
  SEX: Stimulating [Low Volume Gel] | 2.35 (1.05) | 2.58 (1.04)
  SEX: Stimulating [High Volume Gel] | 2.72 (0.85) | 2.66 (0.98)
  SEX: Stimulating [Film] | 1.36 (0.73) | 1.99 (0.92)
  SEX: Messiness [Low Volume Gel] | 1.65 (0.69) | 1.84 (0.70)
  SEX: Messiness [High Volume Gel] | 2.11 (0.81) | 2.18 (0.80)
  SEX: Messiness [Film] | 1.39 (0.49) | 1.32 (0.33)
  SEX: Perceived Leakage [Low Volume Gel] | 2.05 (0.89) | 1.73 (0.57)
  SEX: Perceived Leakage [High Volume Gel] | 2.44 (0.95) | 2.10 (0.77)
  SEX: Perceived Leakage [Film] | 1.48 (0.62) | 1.38 (0.45)
  SEX: Perceived Naturalness [Low Volume Gel] | 3.38 (0.81) | 3.17 (0.95)
  SEX: Perceived Naturalness [High Volume Gel] | 3.44 (0.93) | 3.17 (0.97)
  SEX: Perceived Naturalness [Film] | 2.40 (1.23) | 2.60 (1.42)
  SEX: Perceived Lubricity [Low Volume Gel] | 3.10 (1.20) | 3.15 (1.10)
  SEX: Perceived Lubricity [High Volume Gel] | 3.50 (1.08) | 3.42 (1.05)
  SEX: Perceived Lubricity [Film] | 1.38 (0.63) | 1.63 (0.80)
  SEX: Effortful [Low Volume Gel] | 1.41 (0.59) | 1.53 (0.76)
  SEX: Effortful [High Volume Gel] | 1.17 (0.46) | 1.19 (0.47)
  SEX: Effortful [Film] | 3.08 (1.53) | 2.81 (1.26)
  SEX: Pleasure [Low Volume Gel] | 2.35 (0.97) | 2.88 (0.82)
  SEX: Pleasure [High Volume Gel] | 2.93 (1.04) | 2.92 (1.00)
  SEX: Pleasure [Film] | 1.43 (0.87) | 2.08 (0.90)
  SEX: Perceived Pre-Sex Leakage [Low Volume Gel]: number analyzed (Participants) | 24 | 0
  SEX: Perceived Pre-Sex Leakage [Low Volume Gel] | 2.08 (1.34) |
  SEX: Perceived Pre-Sex Leakage [High Volume Gel]: number analyzed (Participants) | 24 | 0
  SEX: Perceived Pre-Sex Leakage [High Volume Gel] | 2.89 (1.49) |
  SEX: Perceived Pre-Sex Leakage [Film]: number analyzed (Participants) | 24 | 0
  SEX: Perceived Pre-Sex Leakage [Film] | 1.25 (0.72) |
  SEX: Noticeable [Low Volume Gel] | 2.14 (1.00) | 2.54 (1.01)
  SEX: Noticeable [High Volume Gel] | 2.65 (1.29) | 2.89 (1.07)
  SEX: Noticeable [Film] | 1.75 (1.19) | 1.78 (0.78)

ADVERSE EVENTS:
Time Frame: On average, 12 to 16 weeks
Groups:
- Females: Female member of couple enrolled
- Males: Male member of couple enrolled
Arm/Group | Females | Males
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 6/24 | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Females (N=24) | Males (N=24)
Vaginal Dryness (Reproductive system and breast disorders) | 5 (5) | 0 (0)
Pain (vaginal introitus; penis) (Reproductive system and breast disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
User Sensory Perceptions & Experience (USPE) scales adapted and were used for the first time with male sexual partners in Project MIST.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No